CLINICAL TRIAL: NCT05474196
Title: Association Between Driving Transpulmonary Pressure and Extravascular Lung Water in Patients with ARDS
Status: Recruiting | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Tai PHAM, Principal Investigator, Bicetre Hospital
Other Study IDs: 2022-A01289-34
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Intubated patients with the acute respiratory distress syndrome (ARDS) are usually treated with protective ventilation limiting plateau pressure below 30 centimeter of water (cmH2O) and, if possible, a driving pressure under 15 cmH2O. However, these airway pressures might not reflect the actual pressure applied to the lung. Transpulmonary pressure is the difference between airway pressure and pleural pressure, the latter is estimated by the esophageal pressure, and so it better reflects the ventilatory induced lung injury (VILI).

One of the consequences of the VILI is a increase of pulmonary edema and it could be estimated by the extravascular lung water, obtained by trans-pulmonary thermodilution.

So it could exist a link between the driving trans-pulmonary pressure and the extravascular lung water.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory distress syndrome (ARDS)
* Monitoring with a transpulmonary thermodilution device
* Esophageal pressure monitoring

Exclusion Criteria:

* Legal protection measures
* Pregnancy
* Contra-indications of esophageal catheter : esophageal varicose, severe coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intubated in the medical ICU of Bicêtre hospital (Academic hospital), Le Kremlin Bicêtre, France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Association between the transpulmonary driving pressure and the extravascular lung water (EVLW) | From inclusion up to hospital discharge (maximum day 60)
  On the first day of patient's respiratory and hemodynamics monitoring, we will collect transpulmonary driving pressure and extra-vascular lung water values. We will calculate the correlation coefficient linking these two variables to assess if their association.

SECONDARY OUTCOMES:
Association between the transpulmonary driving pressure and the pulmonary vascular permeability index (PVPI) | From inclusion up to hospital discharge (maximum day 60)
  On the first day of patient's respiratory and hemodynamics monitoring, we will collect transpulmonary driving pressure and PVPI values. We will calculate the correlation coefficient linking these two variables to assess if their association.
Correlation between the transpulmonary driving pressure at admission and the ICU-mortality | From inclusion up to hospital discharge (maximum day 60)
  Multivariable analysis of factors associated with ICU mortality, including initial severity, comorbidities, respiratory mechanics covariates, EVLW and pulmonary vascular permeability index (PVPI).
Correlation between the extravascular lung water at admission and the ICU-mortality | From inclusion up to hospital discharge (maximum day 60)
  Multivariable analysis of factors associated with ICU mortality, including initial severity, comorbidities, respiratory mechanics covariates, EVLW and pulmonary vascular permeability index (PVPI).
Influence of position on plateau pressure | From inclusion up to hospital discharge (maximum day 60)
  Plateau pressure will be measured at 0°, 30° and 45° position and we will compare the values to assess if the position impacts this pressure.
Influence of position on plateau pressure on esophageal pressure | From inclusion up to hospital discharge (maximum day 60)
  Esophageal pressure will be measured at 0°, 30° and 45° position and we will compare the values to assess if the position impacts this pressure.
Influence of position on plateau pressure on transpulmonary pressure | From inclusion up to hospital discharge (maximum day 60)
  Transpulmonary pressure will be measured at 0°, 30° and 45° position and we will compare the values to assess if the position impacts this pressure.
Influence of position on plateau pressure on intra-abdominal pressure | From inclusion up to hospital discharge (maximum day 60)
  Intra-abdominal pressure will be measured at 0°, 30° and 45° position and we will compare the values to assess if the position impacts this pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Tài Pham, MD, PhD, Principal Investigator — Hôpital Bicêtre
Locations (1):
- Medical Intensive Care Unit, Bicêtre Hospital, Le Kremlin-Bicêtre, France